CLINICAL TRIAL: NCT00062634
Title: Female Condom Intervention Trial
Brief Title: Education Program to Promote Female Condom Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: HD39118
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: HIV Infections
Keywords: Female condom use; Male condom use; AIDS education; AIDS prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Female condom skills training

SUMMARY:
The female condom offers women a potentially important option for HIV prevention. This study will develop and evaluate a health education program to increase female condom use among ethnically diverse women.

DETAILED DESCRIPTION:
AIDS incidence among women has grown at alarming rates since 1985. Heterosexual contact is now the greatest risk for HIV infection in women. Women in the United States urgently need more options to protect themselves against HIV. Nonetheless, limited prevention efforts have targeted women. The female condom is a potentially important option for HIV prevention in women. However, little research has been conducted to identify effective approaches to promote the female condom as the only female-controlled barrier method available to date. This study will develop a theoretically and empirically based intervention to increase female condom use among ethnically diverse women who engage in multiple sexual partnerships.

The proposed female condom skills training intervention applies social cognitive theory. It also incorporates our extensive previous research that examined female condom acceptability and identified the attitudinal, interpersonal, and sociocultural factors affecting female condom use. The intervention consists of four sessions: 1) individual safer sex education and condom use skills training; 2) group discussion of barriers to female condom use; 3) group condom negotiation skills training; and 4) individual condom use counseling. The efficacy of the intervention will be assessed by comparing it to a control condition intervention that focuses on women's general health issues unrelated to HIV/AIDS. The control condition intervention has four sessions: 1) individual health education; 2) group discussion of women's health problems and related risk behaviors; 3) group discussion of healthy living; and 4) individual health risk reduction counseling.

This study will use a randomized clinical trial design. Study participants will be randomly assigned to one of two conditions: female condom skills training or women's general health promotion. All participants will be interviewed at study entry, 3 months, and 6 months. Attitudinal, psychosexual, and behavioral data will be collected to evaluate the intervention.

ELIGIBILITY:
Inclusion Criteria

* African American, Asian American, Latina, or White
* Two or more male sexual partners in the year prior to study entry
* English speaking

Exclusion Criteria

* Commercial sex workers
* Planning to move within 6 months of study entry
* Allergic to polyurethane, latex, or lubricants

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2003-06; Study Completion 2005-08

PRIMARY OUTCOMES:
percent of sex acts protected by female condoms

SECONDARY OUTCOMES:
percent of sex acts protected by male or female condoms

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hee Choi, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Center for AIDS Prevention Studies, University of California, San Francisco, San Francisco, California, United States